CLINICAL TRIAL: NCT05652764
Title: The Effect of Orem's Self-Care Deficit Theory Based Nursing Interventions on Symptom Management, Care Needs and The Quality of Life of Immunotherapy Treated Cancer Patients
Brief Title: Orem's Self-Care Deficit Theory Based Nursing Interventions for Immunotherapy Treated Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Mevlüde Ergen, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KAEK- 685
Record Dates: First submitted 2022-12-03; First posted 2022-12-15 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Cancer; Nurse's Role; Treatment Side Effects; Quality of Life
Keywords: Cancer Immunotherapy; Treatment Side Effects; Symptom Management; Self-Care Deficiency; Care Needs; Oncology Nursing
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial consisting of two groups: experimental and control.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immuno-SelfCare (Experimental)
  Interventions: Other: Orem's Self-Care Deficit Theory Based Nursing Interventions for Immunotherapy Treated Cancer Patients
- Control Group (No Intervention)

INTERVENTIONS:
Other: Orem's Self-Care Deficit Theory Based Nursing Interventions for Immunotherapy Treated Cancer Patients — In this study, face-to-face patient education, giving patient education booklet, preparation of symptom management card, face-to-face and telephone counseling initiatives were planned to the experimental group.
  Arms: Immuno-SelfCare

SUMMARY:
Objective: The aim of this study was to determine the effects of nursing interventions based on Orem Self-Care Deficiency Theory on symptom management, care needs and quality of life in cancer patients who underwent immunotherapy.

Method: The research was planned as a randomized controlled trial. The research is planned to be carried out in the Medical Oncology unit of the Health Sciences University Antalya Training and Research Hospital. It is planned to be done with 58 patients, 29 experimental and 29 control groups. Based on Orem Self-Care Deficit Theory; face-to-face patient education, giving patient education booklet, preparation of symptom management card, face-to-face and telephone counseling initiatives were planned. Patient Description Form, Supportive Care Needs Scale-Short Form, Memorial Symptom Assessment Scale, European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Scale and Self-Care Strength Scale will be used to collect data.

ELIGIBILITY:
Inclusion Criteria:

* Coming to Antalya Training and Research Hospital Medical Oncology unit for treatment,
* First time taking one of the immune checkpoint inhibitors (Ipilimumab CTLA-4, Pembrolizumab PD-1, Nivolumab PD-1, Atezolizumab PDL-1),
* Speaking and understanding Turkish,
* Being literate,
* 18 Years and older
* With solid tumor,
* No communication barrier
* Being able to communicate by phone
* Individuals who agree to participate in the research.

Exclusion Criteria:

* Patients receiving other cancer treatments in combination with immunotherapy,
* Patients with Eastern Cooperative Oncology Group Performance Scale 4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Symptom on the Memorial Symptom Assessment Scale at week 12 | Baseline and 12th week
  Memorial Symptom Assessment Scale (MSAS): The Memorial Symptom Assessment Scale is a multidimensional self-report questionnaire that evaluates 32 physical and psychological symptoms according to their frequency, severity and distress/bother to the person in the past week.The total score is the average of the responses to the distress scale items and and ranges from 0 to 4 with higher values indicating greater distress experienced from symptoms.
Change from Baseline in Supportive Care Needs on the Supportive Care Needs Scale-Short Form at week 12 | Baseline and 12th week
  Supportive Care Needs Scale-Short Form: The 31-item instrument measures supportive care needs in five domains: health system and information, psychological needs, physical and daily living, patient care and support, and sexual-related. Responses are given on a scale from 1 to 5 where 1 = no help is needed and 5 = high need for help. Total scores range from 31 to 155 and higher scores indicate greater need for help.
Change from Baseline in Self-Care Strength on the Self-Care Strength Scale at week 12 | Baseline and 12th week
  Self-Care Strength Scale: A maximum score of 140 is taken from the scale. The high score obtained from the scale indicates the high level of self-care or self-care ability and power of the individual.
Change from Baseline in Quality of Life Level on the EORTC QLQ-C30 Quality of Life Scale(European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire) at week 12 | Baseline and 12th week
  EORTC QLQ-C30 Quality of Life Scale(European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire): This Scale was developed to measure the quality of life of patients with cancer. It includes 30 questions and three sub-dimensions: General Well-Being, Functional Difficulties, and Symptom Control. The maximum score on the scale is 100, and the minimum is 0. High scores on the functional sub-dimension indicate good/healthy functional status, high scores on the symptom sub-dimension indicate high levels of symptoms and/or problems, and high scores on the global health status/quality of life sub-dimension indicate good quality of life.
Change from Baseline in Adverse Events on the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 for 12 weeks | Baseline,for 12 weeks
  NCI-Common Terminology Criteria for Adverse Events Version 5.0: These algorithms provide support for prescribing the necessary treatment for grade 1 and grade 2 adverse events and for creating special care plans for grade 3 and 4 adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Arikan, Study Director — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No